CLINICAL TRIAL: NCT04280289
Title: CBD Cannabis Extract: Pharmacokinetic Studies
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Mississippi, Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CBD Study 1
Record Dates: First submitted 2020-02-07; First posted 2020-02-21 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Epilepsy
Keywords: CBD; cannabidiol extract; cannabidiol; CBDE; pharmacokinetics
MeSH Terms: conditions — Epilepsy | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: This study is a single center, prospective, Phase I PK trial. A total of 10 healthy subjects will be enrolled into the study. This study will evaluate the pharmacokinetics of CBDE.
  The PK of CBD, 9-tetrahydrocannabinol (THC) and their principal metabolites will be determined after a single CBDE dose delivering 2.5 mg/kg CBD. ). CBDE will be provided in liquid concentration of 50mg/ml in sesame seed oil (SSO).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cannabidiol extract (Experimental): 10 healthy subjects (5 female, 5 male), will be enrolled into the study. Each subject will receive a single CBDE dose delivering 2.5 mg/kg CBD, after consumption of a standardized meal.
  Nine (9mL) of blood for PK analysis, at each of the following timepoints: 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours and 72 hours after the study drug administration.
  Urine will be collected at the following timepoints: Predose, 0-4 hrs, 4-8 hrs, 8-12 hrs, 12-24 hrs, 24-36 hrs, 36-48 hrs, and 48-72 hrs for PK analysis
  Interventions: Drug: cannabidiol extract

INTERVENTIONS:
Drug: cannabidiol extract — The test article "CBD Cannabis Extract Oral Solution" will be manufactured by the University of Mississippi National Center for Natural Products Research (NCNPR) at the Coy Waller Laboratory under FDA Current Good Manufacturing Practices. The drug product, derived from hemp and containing less than 0.3% of Δ9-tetrahydrocannabinol, is no longer a Drug Enforcement Agency (DEA) controlled substance. DEA registrations are not required for the manufacturing, handling or dispensing of these clinical test materials
  Other Names: cannabidiol, CBD

SUMMARY:
The initial goal is to ascertain the pharmacokinetic (PK) profile of CBD (cannabidiol) after a single dose of CBDE (cannabidiol extract), although the plan is to extend these studies to multiple dose administrations in the future, since it is likely that (cannabidiol) and/or its metabolites will show some accumulation. These studies will provide detailed information that will inform the continuation and expansion of CBDE in other research projects.

DETAILED DESCRIPTION:
The objective is to determine the PK profile of CBD(cannabidiol) , its metabolites, and minor phytocannabinoids after single dose administration of CBDE (at 2.5 mg/kg CBD). Attainment of this goal will provide essential information on phytocannabinoid disposition and dosing regimen optimization. To accomplish this objective, the working hypothesis that complex phytochemical mixtures present in full spectrum hemp extracts (FSHEs), as exemplified by CBDE, differ from purified CBD-containing products with regard to PK, will be tested. The approach to testing this working hypothesis will be to use liquid chromatography-mass spectrometry (LC/MS) to both characterize the phytocannabinoid concentration-time profiles following CBDE administration (single and multiple dosing).

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy adults aged 21 to 55 years

Exclusion Criteria:

* Allergy to sesame oil/products

  * Obese: BMI is 35 or higher
  * Smoker (tobacco & marijuana use [smoking or use of oral hemp/CBD products])
  * Currently any taking prescriptions medication(s) [with exception of oral contraceptives] or over-the-counter medications/supplements
  * Consuming botanical/non-botanical dietary supplements (3 days prior to study)
  * Known history of cardiac, liver, kidney or hematological disease, diabetes
  * Autoimmune disorders
  * Known history of Neurologic/Psychiatric disorders
  * Report of an active infection
  * Subject is pregnant or breast-feeding, or is expecting to conceive during the study
  * Subjects of child bearing potential will use (or is currently using) during the study, one of the following acceptable methods of contraception:

Male sterilization (vasectomy) Female sterilization (tubal ligation, hysterectomy) Intrauterine service intrauterine device (IUD) or other implant Oral contraceptive, injectable contraceptive Contraceptive patch/ring Diaphragm Male condom Sponge/spermicide

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of minor phytocannabinoids, and metabolites following single dose administration of Cannabis extract (CBDE) (at 2.5 mg/kg cannabidiol (CBD). | 0- 72 hours
  This study would provide information on differential pharmacokinetics and metabolism of Cannabis extract in normal human volunteers
Urine concentration of minor phytocannabinoids, and metabolites following single dose administration of Cannabis extract (CBDE) (at 2.5 mg/kg cannabidiol (CBD). | 0- 72 hours
  This study would provide information on differential pharmacokinetics and metabolism of Cannabis extract in normal human volunteers

SECONDARY OUTCOMES:
Area-under-the-concentration-time profiles (AUC), and area-under-the moment curve (AUMC), for CBD (cannabidiol) , up to 72 hours after Cannabis extract administration. | 0-72 hours
  This study would provide information on differential pharmacokinetics and metabolism of Cannabis extract in normal human volunteers
Clearance (Cl/F) up to 72 hours after Cannabis extract administration. | 0-72 hours
  This study would provide information on differential pharmacokinetics and metabolism of Cannabis extract in normal human volunteers
Volume of distribution (Vd),up to 72 hours after Cannabis extract administration. | 0-72 hours
  This study would provide information on differential pharmacokinetics and metabolism of Cannabis extract in normal human volunteers
Volume of distribution at steady state (Vdss),up to 72 hours after Cannabis extract administration. | 0-72 hours
  This study would provide information on differential pharmacokinetics and metabolism of Cannabis extract in normal human volunteers.
Terminal elimination rate constant (ke), half-life (t1/2), up to 72 hours after Cannabis extract administration. | 0-72 hours
  This study would provide information on differential pharmacokinetics and metabolism of Cannabis extract in normal human volunteers.
Mean residence time (MRT), up to 72 hours after Cannabis extract administration. | 0-72 hours
  This study would provide information on differential pharmacokinetics and metabolism of Cannabis extract in normal human volunteers.
Maximum serum concentration (Cmax), up to 72 hours after Cannabis extract administration. | 0-72 hours
  This study would provide information on differential pharmacokinetics and metabolism of Cannabis extract in normal human volunteers.
Time to reach Cmax (Tmax), up to 72 hours after Cannabis extract administration. | 0-72 hours
  This study would provide information on differential pharmacokinetics and metabolism of Cannabis extract in normal human volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Bill Gurley, Ph. D., Principal Investigator — Principal Scientist, National Center for Natural Products Research
Locations (1):
- University of Mississippi, University, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolff V, Jouanjus E. Strokes are possible complications of cannabinoids use. Epilepsy Behav. 2017 May;70(Pt B):355-363. doi: 10.1016/j.yebeh.2017.01.031. Epub 2017 Feb 23. PMID 28237318
- [Result] Bonn-Miller MO, Loflin MJE, Thomas BF, Marcu JP, Hyke T, Vandrey R. Labeling Accuracy of Cannabidiol Extracts Sold Online. JAMA. 2017 Nov 7;318(17):1708-1709. doi: 10.1001/jama.2017.11909. PMID 29114823
- [Result] Borchardt D. Hemp cannabis product sales projected to hit $1 billion in 3 years. Forbes 2017, August, 23.
- [Result] Carvalho RK, Andersen ML, Mazaro-Costa R. The effects of cannabidiol on male reproductive system: A literature review. J Appl Toxicol. 2020 Jan;40(1):132-150. doi: 10.1002/jat.3831. Epub 2019 Jul 17. PMID 31313338
- [Result] Devinsky O, Marsh E, Friedman D, Thiele E, Laux L, Sullivan J, Miller I, Flamini R, Wilfong A, Filloux F, Wong M, Tilton N, Bruno P, Bluvstein J, Hedlund J, Kamens R, Maclean J, Nangia S, Singhal NS, Wilson CA, Patel A, Cilio MR. Cannabidiol in patients with treatment-resistant epilepsy: an open-label interventional trial. Lancet Neurol. 2016 Mar;15(3):270-8. doi: 10.1016/S1474-4422(15)00379-8. Epub 2015 Dec 24. PMID 26724101
- [Result] Devinsky O, Cross JH, Laux L, Marsh E, Miller I, Nabbout R, Scheffer IE, Thiele EA, Wright S; Cannabidiol in Dravet Syndrome Study Group. Trial of Cannabidiol for Drug-Resistant Seizures in the Dravet Syndrome. N Engl J Med. 2017 May 25;376(21):2011-2020. doi: 10.1056/NEJMoa1611618. PMID 28538134
- [Result] Devinsky O, Patel AD, Thiele EA, Wong MH, Appleton R, Harden CL, Greenwood S, Morrison G, Sommerville K; GWPCARE1 Part A Study Group. Randomized, dose-ranging safety trial of cannabidiol in Dravet syndrome. Neurology. 2018 Apr 3;90(14):e1204-e1211. doi: 10.1212/WNL.0000000000005254. Epub 2018 Mar 14. PMID 29540584
- [Result] Ewing LE, Skinner CM, Quick CM, Kennon-McGill S, McGill MR, Walker LA, ElSohly MA, Gurley BJ, Koturbash I. Hepatotoxicity of a Cannabidiol-Rich Cannabis Extract in the Mouse Model. Molecules. 2019 Apr 30;24(9):1694. doi: 10.3390/molecules24091694. PMID 31052254
- [Result] Ewing LE, McGill MR, Yee EU, Quick CM, Skinner CM, Kennon-McGill S, Clemens M, Vazquez JH, McCullough SS, Williams DK, Kutanzi KR, Walker LA, ElSohly MA, James LP, Gurley BJ, Koturbash I. Paradoxical Patterns of Sinusoidal Obstruction Syndrome-Like Liver Injury in Aged Female CD-1 Mice Triggered by Cannabidiol-Rich Cannabis Extract and Acetaminophen Co-Administration. Molecules. 2019 Jun 17;24(12):2256. doi: 10.3390/molecules24122256. PMID 31212965
- [Result] Foster BC, Abramovici H, Harris CS. Cannabis and Cannabinoids: Kinetics and Interactions. Am J Med. 2019 Nov;132(11):1266-1270. doi: 10.1016/j.amjmed.2019.05.017. Epub 2019 May 30. PMID 31152723
- [Result] Grof CPL. Cannabis, from plant to pill. Br J Clin Pharmacol. 2018 Nov;84(11):2463-2467. doi: 10.1111/bcp.13618. Epub 2018 May 24. PMID 29701252
- [Result] (Harvey et al; Ujvary and Hanus; Jiang et al; Huestis, etc.1999): CBD is a potent inhibitor of CYP450 isozymes, primarily CYP2C and CYP3A isoforms, in in vitro and animal models
- [Result] Huestis MA, Solimini R, Pichini S, Pacifici R, Carlier J, Busardo FP. Cannabidiol Adverse Effects and Toxicity. Curr Neuropharmacol. 2019;17(10):974-989. doi: 10.2174/1570159X17666190603171901. PMID 31161980
- [Result] H.R.2 - Agriculture Improvement Act of 2018, Public Law No: 115-334, Dec. 20, 2018.
- [Result] McCoy B, Wang L, Zak M, Al-Mehmadi S, Kabir N, Alhadid K, McDonald K, Zhang G, Sharma R, Whitney R, Sinopoli K, Snead OC 3rd. A prospective open-label trial of a CBD/THC cannabis oil in dravet syndrome. Ann Clin Transl Neurol. 2018 Aug 1;5(9):1077-1088. doi: 10.1002/acn3.621. eCollection 2018 Sep. PMID 30250864
- [Result] Morrison G, Crockett J, Blakey G, Sommerville K. A Phase 1, Open-Label, Pharmacokinetic Trial to Investigate Possible Drug-Drug Interactions Between Clobazam, Stiripentol, or Valproate and Cannabidiol in Healthy Subjects. Clin Pharmacol Drug Dev. 2019 Nov;8(8):1009-1031. doi: 10.1002/cpdd.665. Epub 2019 Feb 21. PMID 30791225
- [Result] Pamplona FA, da Silva LR, Coan AC. Corrigendum: Potential Clinical Benefits of CBD-Rich Cannabis Extracts Over Purified CBD in Treatment-Resistant Epilepsy: Observational Data Meta-analysis. Front Neurol. 2019 Jan 10;9:1050. doi: 10.3389/fneur.2018.01050. eCollection 2018. PMID 30687209
- [Result] Personal statement from principal investigator, Dr. John Ingram, Dept. of Pediatrics, University of Mississippi Medical Center on his experience with "Cannabidiol (CBD) Cannabis Extract Oral Solution for Drug Resistant Pediatric Epilepsy (Compassionate Use)," April 18, 2018.
- [Result] Purohit V, Rapaka R, Shurtleff D. Role of cannabinoids in the development of fatty liver (steatosis). AAPS J. 2010 Jun;12(2):233-7. doi: 10.1208/s12248-010-9178-0. Epub 2010 Mar 5. PMID 20204561
- [Result] Russo EB. Beyond Cannabis: Plants and the Endocannabinoid System. Trends Pharmacol Sci. 2016 Jul;37(7):594-605. doi: 10.1016/j.tips.2016.04.005. Epub 2016 May 11. PMID 27179600
- [Result] Russo EB. Taming THC: potential cannabis synergy and phytocannabinoid-terpenoid entourage effects. Br J Pharmacol. 2011 Aug;163(7):1344-64. doi: 10.1111/j.1476-5381.2011.01238.x. PMID 21749363
- [Result] Szaflarski JP, Bebin EM, Cutter G, DeWolfe J, Dure LS, Gaston TE, Kankirawatana P, Liu Y, Singh R, Standaert DG, Thomas AE, Ver Hoef LW; UAB CBD Program. Cannabidiol improves frequency and severity of seizures and reduces adverse events in an open-label add-on prospective study. Epilepsy Behav. 2018 Oct;87:131-136. doi: 10.1016/j.yebeh.2018.07.020. Epub 2018 Aug 9. PMID 30100226
- [Result] Taylor L, Gidal B, Blakey G, Tayo B, Morrison G. A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose, Multiple Dose, and Food Effect Trial of the Safety, Tolerability and Pharmacokinetics of Highly Purified Cannabidiol in Healthy Subjects. CNS Drugs. 2018 Nov;32(11):1053-1067. doi: 10.1007/s40263-018-0578-5. PMID 30374683
- [Result] Taylor L, Crockett J, Tayo B, Morrison G. A Phase 1, Open-Label, Parallel-Group, Single-Dose Trial of the Pharmacokinetics and Safety of Cannabidiol (CBD) in Subjects With Mild to Severe Hepatic Impairment. J Clin Pharmacol. 2019 Aug;59(8):1110-1119. doi: 10.1002/jcph.1412. Epub 2019 Mar 28. PMID 30921490
- [Result] Tzadok M, Uliel-Siboni S, Linder I, Kramer U, Epstein O, Menascu S, Nissenkorn A, Yosef OB, Hyman E, Granot D, Dor M, Lerman-Sagie T, Ben-Zeev B. CBD-enriched medical cannabis for intractable pediatric epilepsy: The current Israeli experience. Seizure. 2016 Feb;35:41-4. doi: 10.1016/j.seizure.2016.01.004. Epub 2016 Jan 6. PMID 26800377
- [Result] Wang YH, Avula B, ElSohly MA, Radwan MM, Wang M, Wanas AS, Mehmedic Z, Khan IA. Quantitative Determination of Delta9-THC, CBG, CBD, Their Acid Precursors and Five Other Neutral Cannabinoids by UHPLC-UV-MS. Planta Med. 2018 Mar;84(4):260-266. doi: 10.1055/s-0043-124873. Epub 2017 Dec 20. PMID 29262425
- See also: US FDA Hearing on Cannabis-Derived Compounds and Products — https://www.fda.gov/media/128592/download